CLINICAL TRIAL: NCT05441501
Title: A Phase 1 Study of JNJ-80038114, a T-Cell Redirecting Agent Targeting Prostate Specific Membrane Antigen (PSMA), for Advanced Stage Prostate Cancer
Brief Title: A Study of JNJ-80038114 in Participants With Advanced Stage Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109209; 80038114PCR1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive JNJ-80038114. The dose levels will be escalated based on the dose limiting toxicities (DLTs) evaluation by the study evaluation team (SET).
  Interventions: Drug: JNJ-80038114
- Part 2: Dose Expansion (Experimental): Participants will receive JNJ-80038114 at the recommended Phase 2 dose (RP2D) determined in Part 1.
  Interventions: Drug: JNJ-80038114

INTERVENTIONS:
Drug: JNJ-80038114 — JNJ-80038114 will be administered.

SUMMARY:
The purpose of this study is to determine recommended phase 2 dose(s) (RP2Ds) of JNJ-80038114 in Part 1 (dose escalation) and to determine the safety at the RP2D(s) in Part 2 (dose expansion).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration-resistant prostate cancer (mCRPC) with confirmed adenocarcinoma of the prostate as defined by Prostate Cancer Working Group 3 (PCWG3)
* Measurable or evaluable disease
* At least 1 prior treatment for mCRPC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ functions as defined by certain laboratory values
* Must sign an informed consent form (ICF)
* Participants must agree to use a highly effective form of birth control as guided by the study doctor

Exclusion Criteria:

* Concurrent anticancer therapy
* Severe or long-lasting side effects related to prior anticancer therapy
* Known allergies to JNJ-80038114 or its excipients
* Brain metastasis or known seizure history
* Significant infections or lung, heart or other medical conditions

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 2: Number of Participants With Adverse Events (AEs) | Up to 2 Years 6 Months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Parts 1 and 2: Number of Participants With AEs by Severity | Up to 2 Years 6 Months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event. Cytokine release syndrome (CRS) and associated neurologic toxicity events will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines.
Part 1: Number of Participants With Dose-Limiting Toxicity (DLT) | Up to 2 Years 6 Months
  Number of participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Serum Concentration of JNJ-80038114 | Up to 2 Years 6 Months
  Serum concentration of JNJ-80038114 will be determined.
Systemic Cytokine Concentrations | Up to 2 Years 6 Months
  Cytokine concentrations will be determined for biomarker assessment.
Serum Prostate Specific Antigen (PSA) Concentration | Up to 2 Years 6 Months
  Serum PSA concentration will be determined.
Number of Participants With Antibodies to JNJ-80038114 | Up to 2 Years 6 Months
  Serum samples will be analyzed for the detection of antibodies to JNJ-80038114 using a validated assay method.
Objective Response Rate (ORR) | Up to 2 Years 6 Months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to Prostate Cancer Working Group 3 (PCWG3) response criteria.
PSA Response Rate | Up to 2 Years 6 Months
  PSA response rate is defined as the percentage of participants with a confirmed decline in PSA of 50 percent (%) or more from baseline.
Duration of Response (DOR) | Up to 2 Years 6 Months
  DOR is defined as the duration from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3 response criteria, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- United States (3):
  - University Of Minnesota, Minneapolis, Minnesota
  - Sidney Kimmel Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
- United Kingdom (3):
  - University College London Hospitals NHSFT, London
  - The Christie NHS Foundation Trust Christie Hospital, Manchester
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Hudson A, Jayaram A, Garmezy B, Zorko NA, Zarrabi KK, Mathews L, Rupnow B, Li M, Ghosh D, Urtishak K, Francis P, Wang SC, Attiyeh E, de Bono J. A phase 1, first-in-human, dose escalation study of JNJ-80038114, a PSMAxCD3 bispecific antibody, in participants with metastatic castration-resistant prostate cancer. Cancer Chemother Pharmacol. 2026 Jan 6;96(1):5. doi: 10.1007/s00280-025-04846-w. PMID 41493473